CLINICAL TRIAL: NCT00904462
Title: A Randomized, Double-Blind, Pilot Study Comparing the Efficacy and Safety of Lidocaine 5% Patch With Placebo in Patients With Pain From Osteoarthritis of the Knee
Brief Title: Pilot Study of Lidocaine 5% Patch Versus Placebo in Patients With Osteoarthritis Pain of the Knee
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sr. Director, Clinical R&D, Endo Pharmaceuticals Inc
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EN3260-001
Record Dates: First submitted 2009-05-15; First posted 2009-05-19 (Estimated); Last update posted 2010-02-10 (Estimated); Status verified 2010-02

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Lidoderm; Lidocaine; Transdermal Patch

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Lidocaine 5% patch (Experimental): Lidocaine 5% patch (Lidoderm®, Endo Pharmaceuticals Inc.), 1⅓ patches applied on each affected knee once every 24 hours
  Interventions: Drug: Lidoderm
- Placebo patch (Placebo Comparator): Matching placebo patch, 1⅓ patches applied on each affected knee once every 24 hours
  Interventions: Drug: Placebo patch

INTERVENTIONS:
Drug: Lidoderm — Eligible patients were randomly allocated to receive one of two treatments for 12 weeks: lidocaine 5% patch or matching placebo patch.
  Other Names: Lidocaine 5% patch
  Arms: Lidocaine 5% patch
Drug: Placebo patch — Eligible patients were randomly allocated to receive one of two treatments for 12 weeks: lidocaine 5% patch or matching placebo patch.
  Arms: Placebo patch

SUMMARY:
Patients with unilateral or bilateral osteoarthritis (OA) of the knee participated in a Phase II clinical trial to assess the efficacy of lidocaine 5% patch compared with placebo in the treatment of pain from OA of the knee.

ELIGIBILITY:
Key Inclusion Criteria:

1. Had unilateral or bilateral OA of the knee diagnosed according to the American College of Rheumatology (ACR) criteria based on clinical and radiographic evidence (presence of osteophytes on x-ray and written evaluation) of OA
2. Had functional capacity class rating of I, II, or III according to ACR classification
3. Had normal 12-lead electrocardiogram (ECG) without any clinically significant abnormalities in heart rate, rhythm, or conduction
4. Had discontinued use of all analgesic medications (including over-the-counter [OTC] analgesics) prior to randomization (patients were allowed limited use of analgesic medications for non study pain
5. At baseline visit, patients were randomized to double-blind treatment if they had an average pain intensity rating for the index joint of 6 or greater (on a 0 to 10 scale) for at least 3 days out of the 5 consecutive days immediately prior to the baseline visit; 0 is defined as "no pain" and 10 is defined as "pain as bad as ever imagined" as measured by Question 5 of the BPI and recorded in a diary
6. At baseline visit, patients were randomized to double-blind treatment if they had, at the baseline visit, an OA severity score for the index joint of 7 or greater on a composite scale of 0 to 24 as measured by the Index of Severity for Osteoarthrosis of the Knee

Key Exclusion Criteria:

1. Had been diagnosed with inflammatory arthritis, gout, pseudo-gout or Paget's disease that in the investigator's opinion would have interfered with the assessment of pain and other symptoms of OA
2. Had serious medical conditions requiring daily medications, such as anticonvulsants and tricyclic antidepressants, that could have confounded study results
3. Had any other clinically significant joint disease or prior joint replacement surgery at the index joint
4. Had severe renal insufficiency (creatinine clearance of <30 mL/min)
5. Had moderate or greater hepatic impairment
6. Were taking analgesic medications, glucosamine, or chondroitin that could not be discontinued during the study. Patients taking these medications prior to the study were required to discontinue use for the duration of the study. Patients using opioid analgesics at study entry were required to taper off these medications.
7. Were taking long-acting opioids or opioids that could not be discontinued over the first 5 days of the placebo run-in period.
8. Were using lidocaine-containing product that could not be discontinued during the study
9. Had previously failed treatment with Lidoderm analgesic patch for OA
10. Had recently received either a corticosteroid injection (within 8 weeks) or hyaluronic acid (within 6 months) of study entry
11. Were unable to discontinue use of topical drugs applied to the knee
12. Were taking class I anti-arrhythmic drugs (e.g. mexiletine, tocainide)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2004-08; Primary Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities (WOMAC) OA Index | Visit: V2(Day 0), V3(Day 14), V4(Day 28), V5(Day 42), V6(Day 56), V7/EOS(Day 84)
Pain intensity and pain relief (BPI Questions 3, 4, 5, 6, and 8) | Visit: V2(Day 0), V3(Day 14), V4(Day 28), V5(Day 42), V6(Day 56), V7/EOS(Day 84)
Pain Quality Assessment Scale (PQAS) | Visit: V2(Day 0), V3(Day 14), V4(Day 28), V5(Day 42), V6(Day 56), V7/EOS(Day 84)
Patient-rated and Investigator-rated Global Impression of Change in OA pain (categorical scale) | Visit: V2(Day 0), V3(Day 14), V4(Day 28), V5(Day 42), V6(Day 56), V7/EOS(Day 84)
Patient-rated and Investigator-rated Global Assessment of Treatment Satisfaction (categorical scale) | Visit: V2(Day 0), V3(Day 14), V4(Day 28), V5(Day 42), V6(Day 56), V7/EOS(Day 84)

SECONDARY OUTCOMES:
QoL: Pain interference on activities of daily living using Question 9 of the BPI | Visit: V2(Day 0), V3(Day 14), V4(Day 28), V5(Day 42), V6(Day 56), V7/EOS(Day 84)
QoL: Beck Depression Inventory (BDI) | Visit: V2(Day 0), V3(Day 14), V4(Day 28), V5(Day 42), V6(Day 56), V7/EOS(Day 84)
Quality of Sleep (QOS) | Visit: V2(Day 0), V3(Day 14), V4(Day 28), V5(Day 42), V6(Day 56), V7/EOS(Day 84)
Safety assessments included AEs, dermal assessments, clinical laboratory tests (including urinalysis), vital sign measurements, physical examination results, and plasma lidocaine concentrations | Visit: V2(Day 0), V3(Day 14), V4(Day 28), V5(Day 42), V6(Day 56), V7/EOS(Day 84)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Endo Pharmaceuticals
Locations (24):
- United States (24):
  - Birmingham, Alabama
  - Hueytown, Alabama
  - Tallassee, Alabama
  - Phoenix, Arizona
  - Boulder, Colorado
  - DeLand, Florida
  - Largo, Florida
  - Palm Harbor, Florida
  - St. Petersburg, Florida
  - Chicago, Illinois
  - Springfield, Illinois
  - Wheaton, Maryland
  - Peabody, Massachusetts
  - Bingham Farms, Michigan
  - Reno, Nevada
  - Berlin, New Jersey
  - Dayton, Ohio
  - Oklahoma City, Oklahoma
  - Duncansville, Pennsylvania
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
  - Bartlett, Tennessee
  - Cordova, Tennessee
  - Memphis, Tennessee